CLINICAL TRIAL: NCT00573703
Title: A Comparison Between Laparoscopic Burch Colposuspension and Transobturatory Tape (TOT) for the Treatment of Female Urinary Stress Incontinence
Brief Title: Laparoscopic Burch Colposuspension Versus Transobturatory Tape for the Treatment of Female Urinary Stress Incontinence
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02/2007
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Laparoscopic Burch colposuspension; Stress incontinence; Surgery; TOT; Treatment; Predominant or genuine stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator)
  Interventions: Procedure: Laparoscopic Burch colposuspension
- Group B (Experimental)
  Interventions: Procedure: Transobturator tape procedure

INTERVENTIONS:
Procedure: Laparoscopic Burch colposuspension — Lapaparoscopic approach. One or two nonadsorbable sutures are placed at the level of the midurethra without penetrating the vaginal mucosa and fixed to Cooper's ligament with a tension free knotting technique.
  Arms: Group A
Procedure: Transobturator tape procedure — Small incision sites in the vagina and in the femoral/pelvic fold. Bilateral transobturator insertion of mesh by means of needle. Application of resorbable tensioning suture that maintains the mesh and enables fine adjustments in mesh tension during the procedure and in the immediate postoperative period.
  Arms: Group B

SUMMARY:
Transobturatory tape (TOT) procedure is a minimally invasive approach to urinary stress incontinence owing to the category of the sling-adopting procedures. Its efficacy and safety, also in comparison with similar procedures have been demonstrated. The benefits of the sling- adopting procedures in comparison to laparoscopic Burch colposuspension, which has been considered as the gold standard treatment, have been showed. But these comparisons did not included the TOT procedure in the experimental arms. Based on this considerations the aim of this trial will be to compare TOT and laparoscopic Burch colposuspension in women with urinary stress incontinence.

DETAILED DESCRIPTION:
Women with predominant and genuine stress urinary incontinence will be enrolled and randomized in two groups (groups A and B). Patients of group A will be treated with laparoscopic Burch colposuspension, whereas patients of group B will be treated with TOT procedure.

All patients eligible will undergo baseline assessment consisting of anthropometric, clinical, hormonal, urodynamic, and ultrasonographic evaluations. During the study, the surgical outcomes, the clinical subjective and objective efficacy data, and the adverse experiences will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Predominant or genuine stress urinary incontinence by self report,examination and test
* Urethral hypermobility
* Eligible for both surgical procedures
* Ambulatory

Exclusion Criteria:

* Pregnancy
* <12 months post-partum
* Systemic disease and/or drugs known to affect bladder function
* Current chemotherapy or radiation therapy
* Urethral diverticulum, augmentation cytoplasty, or artificial sphincter
* Recent pelvic surgery
* Severe genuine stress incontinence (loss of urine with minimal physical activity) with associated prolapse equal to or more than second degree
* Previous pelvic or anti-incontinence surgery
* History of severe abdominopelvic infections
* Known extensive abdominopelvic adhesions
* Detrusor instability and/or intrinsic sphincter dysfunction
* Other gynaecologic pathologies (eg, fibroids, ovarian cysts)
* BMI >30

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Objective/subjective symptoms improvements | 12 months

SECONDARY OUTCOMES:
Intra-operative complication rate | one day
Postoperative complications rate | 12 months
Failure rate | 12 months
Recurrence rate | 12 months
Quality of life | 12 months
Sexual function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Fulvio Zullo, MD, Study Chair — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Catanzaro, Italy